CLINICAL TRIAL: NCT02424058
Title: The Investigation of the Sagittal Thoracic Spinal Curvature and Mobility in Subjects With and Without Chronic Neck Pain: Cut-off Points and Pain Relationship
Brief Title: The Investigation of Thoracic Spinal Curvature and Mobility in Subjects With and Without Neck Pain: Cut-off Points
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seyda TOPRAK CELENAY, Assistant Professor, PT, PhD, Ataturk Training and Research Hospital
Other Study IDs: 2015-56/32
Record Dates: First submitted 2015-04-12; First posted 2015-04-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Control

GROUPS / COHORTS (2):
- Neck pain: Patients aged between 18 and 65 years with persistent neck pain for more than 3 months
  Interventions: Device: Spinal Mouse® measurement; Behavioral: Neck pain intensity measurement
- Healthy: Acceptance to participate in the study, no previous neck oain (lifetime-to-date), no spinal surgery or deformity, and no radiological abnormalities detected
  Interventions: Device: Spinal Mouse® measurement

INTERVENTIONS:
Device: Spinal Mouse® measurement — The sagittal thoracic spinal curvature and mobility of all participants were assessed with Spinal Mouse® (Idiag, Fehraltorf, Switzerland) in standing position.
Behavioral: Neck pain intensity measurement — The neck pain intensity of the patients was questioned by Visual Analogue Scale
  Groups: Neck pain

SUMMARY:
The purpose of this study is to investigate the sagittal thoracic spinal curvature and mobility in subjects with and without chronic neck pain, cut-off points and pain relationship

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years with persistent neck pain for more than 3 months
* The inclusion criteria for the control group included acceptance to participate in the study, no previous neck pain (lifetime-to-date), no spinal surgery or deformity, and no radiological abnormalities detected

Exclusion Criteria:

* Prior history of injury or surgery relating to spine, spinal deformity, neurological symptoms or signs, radiological abnormalities indicating cervical radiculopathy or myelopathy, prior history of other spinal disorder such as low back pain, active intervention in the last 3 months including drug therapy or physiotherapy, malignancy, systemic pathology including any rheumatologic disease and osteoporosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Chronic neck pain and heatlhy subjects
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Thoracic curvature, as measured by Spinal Mouse® | participants will be followed for the duration of hospital stay, an expected average of one year

SECONDARY OUTCOMES:
Pain, as measured by Visual Analog Scale | participants will be followed for the duration of hospital stay, an expected average of one year
Thoracic mobility, as measured by Spinal Mouse® | participants will be followed for the duration of hospital stay, an expected average of one year

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk Training and Research Hospital, Ankara, Cankaya, Turkey (Türkiye)

REFERENCES:
- [Result] Lau KT, Cheung KY, Chan KB, Chan MH, Lo KY, Chiu TT. Relationships between sagittal postures of thoracic and cervical spine, presence of neck pain, neck pain severity and disability. Man Ther. 2010 Oct;15(5):457-62. doi: 10.1016/j.math.2010.03.009. PMID 20430685
- [Result] Nejati P, Lotfian S, Moezy A, Moezy A, Nejati M. The relationship of forward head posture and rounded shoulders with neck pain in Iranian office workers. Med J Islam Repub Iran. 2014 May 3;28:26. eCollection 2014. PMID 25250268
- [Result] Tsunoda D, Iizuka Y, Iizuka H, Nishinome M, Kobayashi R, Ara T, Yamamoto A, Takagishi K. Associations between neck and shoulder pain (called katakori in Japanese) and sagittal spinal alignment parameters among the general population. J Orthop Sci. 2013 Mar;18(2):216-9. doi: 10.1007/s00776-012-0341-6. Epub 2012 Dec 12. PMID 23232803